CLINICAL TRIAL: NCT05019690
Title: Apatinib Mesylate Combined with Albumin-bound Paclitaxel for Second-line Treatment of Advanced Triple Negative Breast Cancer:a Single-arm,exploratory Clinical Study
Brief Title: Apatinib Combined with Albumin-Bound Paclitaxel for Treatment of Advanced Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-B02
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Triple Negative Breast Cancer
MeSH Terms: interventions — apatinib; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib Combined With Albumin-Bound Paclitaxel (Experimental): Participants will receive apatinib combined with albumin-bound paclitaxel until predefined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Apatinib Mesylate; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Apatinib Mesylate — Subjects receive Apatinib orally, Dosage form: tablet, Strength: 250 mg/tablet,QD,Q3W
  Other Names: apatinib
Drug: Albumin-Bound Paclitaxel — Subjects receive Albumin-Bound Paclitaxel,ivgtt, Strength: 125 mg/m^2,d1、7、15,Q3W
  Other Names: albumin paclitaxel

SUMMARY:
This study is a single-arm,exploratory clinical study, to evaluate the effectiveness and safety of apatinib mesylate combined with albumin-bound paclitaxel for second-line treatment of advanced triple negative breast cancer.

DETAILED DESCRIPTION:
This is a exploratory, single-arm, open-label trial. The investigator's primary purpose is to explore that PFS and safety of apatinib combined with albumin-bound paclitaxel for treatment of advanced triple negative breast cancer.

In treatment period, patients will be administrated apatinib plus albumin-bound paclitaxel, every 21 days for 1 cycle, until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1.Volunteered to participate in the study, signed the informed consent form. 2.Aged 18-75 years,female. 3.Histologically or pathologically confirmed advanced triple-negative breast cancer that meets the following criteria:

  1. Primary tumor stage determined by standard evaluation methods: CT0-4 /N0-3/M1;
  2. Pathologically confirmed breast cancer with negative HER2 expression, defined as < 10% immunoreactive cells with an IHC score of + or -,or in situ hybridization (ISH) resulting in no HER2 gene amplification (RATIO of HER2 gene signal to centromeric 17 signal < 2.0 and HER2 gene copy number/cell < 4.0);
  3. Negative hormone receptor status (ER and PgR) is known, which is defined as < 1% detected by immunohistochemistry;
  4. A previous systemic therapy, including anthracyclines, for recurrence/metastasis.

  4.With measurable lesions,according to Response Evaluation Criteria In Solid Tumors Version 1.1.

  5.Patients must have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale.

  6.Life expectancy ≥12 weeks. 7.No prior treatment with apatinib or albumin paclitaxel, except in neoadjuvant or adjuvant therapy.

  8.Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥80g/L (without blood transfusion during 14 days); a leucopenia count of ≥3.0×109/L; a platelet count of ≥90×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.

  9.Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug.

Exclusion Criteria:

* 1.Pregnant or lactating women. 2.Previous or coexisting malignancies, unless they are basal cell carcinoma of the skin, superficial bladder carcinoma, squamous cell carcinoma of the skin, cervical carcinoma in situ, or other cancers in situ that have achieved complete remission at least 5 years prior to screening and that do not require or are expected to require additional treatment during the study.

  3.Patients with consciousness disorder or unable to cooperate with treatment, with mental illness or metastasis of central nervous system.

  4. Patients who have participated in other clinical trials in the past three months.

  5. Previous treatment with apatinib or other vaso-targeting drugs and other small-molecule tyrosine kinase inhibitors.

  6. Received any targeted treatment before enrollment, including but not limited to the following: surgical treatment, chemotherapy, radiation therapy, targeted therapy, etc.

  7. Within 3 months before treatment, esophageal (fundus) varices were ruptured and bleeding, intestinal obstruction and gastrointestinal perforation.

  8. The subject has clinical symptoms of cancerous ascites or pleural effusion. 9. Subjects have active infection or unexplained fever ≥38.5℃ within 7 days before enrollment.

  10. Severe liver, kidney, heart, lung, brain and other major organ failure. 11. Patients with hypertension who cannot be reduced to the normal range after antihypertensive drug therapy (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg).

  12. Past or present idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, tissue pneumonia (e.g., bronchitis, angiitis oblitans), drug pneumonia, or screening CT with active pneumonia.

  13. Patients with abnormal coagulation (INR > 1.5 or PROthrombin time (PT) > ULN+4 SEC), who are prone to bleeding, or who are receiving thrombolytic or anticoagulant therapy, are permitted to receive low-dose low-molecular heparin or oral aspirin procoagulant therapy during the trial.

  14. Have cardiac clinical symptoms or disease that are not well controlled, e.g. :(1) nyha grade 2 Above heart failure;(2) Unstable angina;(3) Myocardial infarction occurred within 1 year;(4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;(5) QTc > 470ms.

  15. Patients with positive protein urine (urine protein test of 2+ or above, or 24 h urine protein quantification > 1.0g).

  16. Inability to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption.

  17. Overactivity/venous thrombosis events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months before enrollment.

  18. A history of hereditary or acquired bleeding or coagulation disorders.Within 3 months before enrollment, patients with clinically significant bleeding symptoms or a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.

  19. According to the investigator's judgment, the subjects have other factors that may lead to the forced termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which may affect the safety of the subjects or the data collection, etc.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) | From enrollment to 12 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to 24 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Objective response rate(ORR) | From enrollment to 12 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Disease control rate(DCR) | From enrollment to 12 month
  DCR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR or SD. DCR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR or SD to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The DCR will be reported by percentage with each arms and appropriate confidence intervals.
  [Time Frame: From enrollment to 12 month]

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China